CLINICAL TRIAL: NCT03719794
Title: Probiotics for Vascular Inflammation in Metabolic Syndrome (PROMISE): a 12-Week Pilot Study, Randomized,Double-Blinded, Placebo-Controlled Trial
Brief Title: Probiotics for Vascular Inflammation in Metabolic Syndrome
Acronym: PROMISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2016-2038
Record Dates: First submitted 2018-09-12; First posted 2018-10-25 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics arm (Active Comparator): The active comparator arm will be of a 12-week probiotic supplement regimen (one capsule daily, containing 20 x 109 CFU of Bifidobacterium animalis ssp. Lactis Lafti®B94 and Lactobacillus plantarum R1012)
  Interventions: Dietary Supplement: Probiotic supplement
- Placebo arm (Placebo Comparator): The placebo comparator arm will be of a 12-week placebo supplement regimen.
  Interventions: Dietary Supplement: Placebo supplement

INTERVENTIONS:
Dietary Supplement: Probiotic supplement — Probiotic supplement once daily (xyz) for 12 weeks
  Arms: Probiotics arm
Dietary Supplement: Placebo supplement — Placebo supplement once daily for 12 weeks
  Arms: Placebo arm

SUMMARY:
Subjects with metabolic syndrome are known to possess chronic low-level inflammation. Furthermore, such individuals are at risk of developing atherosclerosis in coronary and other vascular beds. In particular, subjects with metabolic syndrome, prediabetes and type II diabetes mellitus were shown to possess vascular inflammation in carotid atherosclerosis as demonstrated using FDG-PET. In the current pilot proposal, the investigators wish to study the impact of 3-month probiotic supplementation on vascular and systemic inflammation in subjects with metabolic syndrome in the context of a randomized, placebo-controlled, pilot trial.

ELIGIBILITY:
Inclusion Criteria:

* Male and female age > 50 years
* Presence of MetS as defined according to recent updated criteria (13): Presence of at least three of five criteria, namely abdominal obesity (waist circumference cut-off) depending on the recently published ethnic-based variations (14), triglycerides > 1.70 mmol/l, decreased HDL-cholesterol (< 1.0 mmol/l in men and < 1.3 mmol/l in women), systolic blood pressure > 130 mmHg or diastolic blood pressure > 85 mmHg, and FPG > 5.6 mmol/l.
* Willingness to complete questionnaires, records, and diaries associated with the study and to complete all clinic visits.
* Willingness to discontinue consumption of fermented foods or probiotics (e.g. yoghourts, with live, active cultures or supplements).
* Able to provide informed consent.

Exclusion Criteria:

* Concurrent consumption of fermented foods or probiotics (e.g. yoghourts, with live, active cultures or supplements). Subjects will be eligible for participation, however, after a two-week washout period
* Overt or documented vascular disease (coronary heart disease, cerebrovascular disease, or peripheral vascular disease).
* Participants suffering from dementia (mini mental state examination) or depression (geriatric depression scale).
* Concurrent statin therapy. (Statins have been shown to reduce vascular inflammation as measured by FDG-PET-see section 9.1).
* Color blind
* Concurrent antibiotic therapy. However, screened participants would be eligible to participate two weeks after completing their course of antibiotics (wash-out period).
* Known to be pregnant or breast-feeding or planning on becoming pregnant in the next 18 months.
* Women of childbearing potential not using effective contraception. Acceptable methods of birth control includes:
* Hormonal contraceptives including combined oral contraceptives, hormone birth control patch, vaginal contraceptive ring, injectable contraceptives, or hormonal implants;
* Intrauterine devices (IUD) or Intrauterine system (IUS);
* Tubal ligation;
* Vasectomy of partner;
* Double barrier method (use of physical barrier by both partners, e.g. male condom and diaphragm, male condom and cervical cap).
* Positive pregnancy test in women of childbearing potential.
* Allergy to milk, soy, or yeast.
* Use of another investigational product within 3 months of the screening visit.
* Claustrophobia
* Patient with pacemaker
* Patient with BMI greater than 40 kg/m2
* Immune disorder.
* Drug and alcohol abuse
* Current use of NSAIDs
* Liver and kidney disorders
* Bleeding/blood disorder

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome is to evaluate the change on vascular inflammation (measured by FDG-PET), so as to test the hypothesis that probiotic treatment reduces vascular inflammation in comparison to placebo. | At baseline and following 12 weeks of probiotic supplementation or placebo.
  PET-CT scan of the carotid arteries and ascending thoracic aorta will be performed 2 hours post I.V. The participant will be injected with 18F-FDG.

SECONDARY OUTCOMES:
Mesure of High-sensitivity C-reactive protein (hs-CRP) a systemic inflammatory marker. | At baseline and following 12 weeks of probiotic supplementation or placebo.
  Change with hs-CRP
Mesure of Tumor necrosis factor alpha (TNF-α) a systemic inflammatory marker. | At baseline and following 12 weeks of probiotic supplementation or placebo.
  Change with TNF-α
Mesure of Matrix metallopeptidase 9 (MMP-9) | At baseline and following 12 weeks of probiotic supplementation or placebo.
  Change with MMP-9
Cognitive function at rest by a standard pen-paper battery test. | At baseline and following 12 weeks of probiotic supplementation or placebo.
  Cognitive functions will be measured at rest with a pen-paper battery test by a neuropsychologist. The investigators will measure change of score to the cognitive tests.
Intestinal microbiota community composition | At baseline and following 12 weeks of probiotic supplementation or placebo.
  To evaluate the impact on intestinal microbiota community composition

OTHER OUTCOMES:
Mesure of blood fasting glucose | At baseline and following 12 weeks of probiotic supplementation or placebo.
  Change in fasting glucose
Mesure of blood Serum lipids | At baseline and following 12 weeks of probiotic supplementation or placebo.
  Change in serum lipids

CONTACTS AND LOCATIONS:
Overall Officials: Anil Nigam, MD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Cardiovascular Prevention and Rehabilitation Center, Montreal, Quebec, Canada